CLINICAL TRIAL: NCT03320226
Title: A Study of the Effect of Probiotics on Gastrointestinal Function During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1028059
Record Dates: First submitted 2017-10-11; First posted 2017-10-25 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Pregnancy Early; Nausea Gravidarum; Vomiting of Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic 10 (Nature's Bounty) (Other): The suggested dose will be two (2) pills of Probiotic 10 (Nature's Bounty) after dinner daily. Subjects will be asked to take probiotics for six (6) days after providing baseline fecal specimen. Subjects will self-report their daily GI function including the frequency of nausea, vomiting, and bowel movement(s). Then, the subjects will stop taking probiotics for two (2) days and resume taking probiotics for another six (6) days. This six (6)-day on and two (2)- day off cycle is repeated two (2) times.
  Interventions: Dietary Supplement: Probiotic 10 (Nature's Bounty)

INTERVENTIONS:
Dietary Supplement: Probiotic 10 (Nature's Bounty) — The Probiotic 10 (Nature's Bounty) that contains 20 billion live cultures of Lactobacillus plantarum 299v (Lp299v®), Lactobacillus bulgaricus Lb-87, Lactobacillus paracasei DSM 13434, Lactobacillus plantarum DSM 15312, Lactobacillus salivarius Ls-33, Lactobacillus brevis Lbr-35, Lactobacillus acidophilus La-14, Bifidobacterium lactis Bl-04, Lactobacillus paracasei Lpc-37, Lactobacillus casei Lc-11, which are under Lactobacillus and Bifidobacterium.

SUMMARY:
The purpose as well as the aim of this project is to understand the effect of probiotics on gastrointestinal (GI) dysfunction such as nausea, vomiting, and constipation that are found during the first and second trimesters of pregnancy.

The primary objective of this project is to uncover whether probiotics have an effect on GI functional disorders.

The secondary objective is to identify the microbiota associated with probiotic intake.

The tested hypothesis is that gut microbiota influences the GI functions and may influence constipation, nausea, and vomiting during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* First and second trimester healthy or low risk pregnant women who report gastrointestinal disorders such as nausea, vomiting, and constipation

Definition of healthy or low risk pregnant women:

* Systolic blood pressure < 140 mmHg and diastolic blood pressure < 90 mmHg
* Hemoglobin ≥ 10.0 g/dL
* Have immunity against rubella (German measles)
* HIV negative
* Urine test shows no sign of kidney or urinary tract infection

  * 27 weeks 6 days gestation or less with confirmed fetal heart beat
  * Pregnant women age 18 and older

Exclusion Criteria:

* High risk pregnant women who have existing health conditions such as high blood pressure, Type 1 diabetes, HIV positive, or are infected with Hepatitis B, Syphilis, or other sexually transmitted diseases
* Pregnant women who have multiple gestations or a history of recurrent miscarriages (more than two consecutive miscarriages)
* Had prior bariatric surgery
* Conceived through IVF program
* Pregnant women who have had severe weight loss (more than 5 pounds) during pregnancy. [Note: Mild weight loss (2-3 pounds) due to nausea, vomiting, or loss of appetite is considered normal.]
* Medical history of irritable bowel syndrome or other non-pregnancy related GI dysfunction/disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — First and second trimester healthy or low risk pregnant women who report gastrointestinal disorders such as nausea, vomiting, and constipation.
Enrollment: 39 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Number of vomiting and nausea per day | 16 days following baseline fecal sample collection
  Using scale of 1-5, quantify the seriousness of sick to the stomach, dry heaves, fatigue, lack of energy, and feeling blue.

SECONDARY OUTCOMES:
The relative quantity of gut bacteria at phylum, family, and species level when patients take or do not take Probiotic-10. | 16 days following baseline fecal sample collection
  To receive at least six (6) analyzable fecal specimens including one prior to taking probiotics from 33 subjects to identify the microbiota associated with probiotic intake.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided